CLINICAL TRIAL: NCT04708652
Title: Relationship Between Neonatal Cerebral Blood Flow Measures and the Neurobehavioral and Handedness Outcomes in Term and Preterm Adolescents
Brief Title: Neonatal Cerebral Blood Flow and the Neurobehavioral and Handedness Outcomes in Term and Preterm Adolescents
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202004122RINC
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Preterm Children
Keywords: handedness; neonatal cerebral blood flow; neurodevelopment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preterm children: Our previous intervention study enrolled 178 VLBW (birth body weight less than 1,500 gm) preterm children who were born or admitted at the National Taiwan University Hospital, the Mackay Memorial Hospital and Taipei City Hospital, Branch for Women and Children in Taipei, Taiwan, during the time period of 2006 to 2008. No any intervention was conducted, just the observation.
  Interventions: Other: No intervention
- term children: Our previous intervention study enrolled 62 term children who were born or admitted at the National Taiwan University Hospital, the Mackay Memorial Hospital and Taipei City Hospital, Branch for Women and Children in Taipei, Taiwan, during the time period of 2006 to 2008. No any intervention was conducted, just the observation.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The results will provide insightful information to understand the process of neural development and the predictive value of early cerebral blood flow measures on longitudinal neurodevelopment and handedness outcomes in preterm and term adolescents. The findings also contribute to the understanding of effectiveness of early intervention on long-term neurodevelopmental outcome in preterm children at adolescence.

Our study has three hypotheses as below:

1. The preterm intervention group have higher neuromotor scores, lower behavioral problem scores and higher incidence of right-handedness than the preterm control group.
2. The preterm intervention group have comparable neuromotor scores, behavioral problem scores and incidence of right-handedness than the term adolescents.
3. The neonatal cerebral blood flow velocity asymmetry measures are significantly associated with the infant, preschool, school and adolescent neurodevelopment and handedness outcomes in preterm children with very low birth weight and term children.

DETAILED DESCRIPTION:
The term and preterm children have previously been administered Cranial Doppler Ultrasound and neurobehavioral assessment at term age, and neurodevelopmental assessment in the neonatal period, infancy, preschool and school age (Bayley Scales of Infant and Toddler Development-3rd edition, Movement Assessment Battery for Children-2nd Edition, Child Behavior Check List/4-18, Wechsler Pre-School and Primary Scales of Intelligence-Revised, and Developmental Test of Visual-Motor Integration - 6th Edition).

All families will be contacted via phone call and mail to participate in this study. Children and their parents will be examined for child neuromotor development, handedness and behavior when the children reach 12-14 years of age. All measures will be conducted at the Infant Motor Development Laboratory, School of Physical Therapy, National Taiwan University. The outcome measures in this study will consist of the growth (weight and height), neuromotor function (Movement Assessment Battery for Children-2nd Edition), handedness (Edinburgh Handedness Inventory) and behavior (child report and parent report of Child Behavior Check List for Ages 4-18 Years).

ELIGIBILITY:
Inclusion Criteria:

Joined our previous study

* preterm group: (1) birth weight <1,500 g; (2) gestational age <37 weeks;
* term group: (1) birth weight >2,500 g; (2) gestation age within 38 and 42 weeks; (3) intrauterine growth status as appropriate for gestational age.

Exclusion Criteria:

* Severe neonatal diseases included major neurologic abnormalities, necrotizing enterocolitis, and severe cardiopulmonary disease and major congenital abnormality.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study extends our previous intervention research. The current study will recruit them for a follow up of their neuromotor development, handedness and behavior outcome after entering junior high school at 12-14 years of age. Our previous intervention study enrolled 178 VLBW preterm children and 62 term children who were born or admitted at the National Taiwan University Hospital, the Mackay Memorial Hospital and Taipei City Hospital, Branch for Women and Children in Taipei, Taiwan, during the time period of 2006 to 2008.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Movement Assessment Battery for Children- 2nd Edition | at age 12-14
  assess movement, <5th percentile categorized as coordinated impairment; 5th-15th percentile categorized as borderline suspicious coordinated impairment; >15th percentile categorized as normal.
Edinburgh Handedness Inventory | at age 12-14
  questionnaire, the assessment of the handedness, not scoring system, not relation to good or bad.
Child Behavior Check List for Ages 4 to 18 Years | at age 12-14
  questionnaire, the assessment of the child behavior, not scoring system, not relation to good or bad.
Neonatal Cranial Doppler Ultrasound | at birth (previous data)
  Cerebral blood flow velocity of the bilateral middle cerebral arteries

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chieh Chou, MD; PhD., Principal Investigator — Department of Pediatrics, National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No